CLINICAL TRIAL: NCT02564731
Title: Prognosis of Bronchiectasis in Children--A Multicenter Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baoping XU (Other)
Collaborators: Wuhan women and children's health care center (Unknown); Children's Hospital of Chongqing Medical University (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Changchun Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); Jiangxi Province Children's Hospital (Other); Shanghai Children's Medical Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Tianjin Children's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Children's Hospital of Fudan University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Other Study IDs: BCHlung003
Record Dates: First submitted 2015-09-14; First posted 2015-10-01 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Bronchiectasis
Keywords: children; prognosis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective cohort study is designed to observe of the effect of intervention therapy on the long-term prognosis of children with bronchiectasis. The main purpose of the study was to evaluate the degree of deterioration of lung function, to observe and compare the quality of life, the time of pulmonary exacerbation, and the changes of lung image.

DETAILED DESCRIPTION:
All enrolled patients are followed up for half a year, 1 years, 2 years, 3 years, 4 years, 5 years, while observation of pulmonary function, symptoms, signs, quality of life, the times of acute pulmonary exacerbation, and the changes of lung image are performed.

ELIGIBILITY:
Inclusion Criteria:A included patient must be coincident at least one point of the four items of high-resolution computed tomography (HRCT) manifestations.

* Internal bronchial diameter greater than the accompanying pulmonary artery.
* lack of bronchial tapering
* bronchi visible in the peripheral 1cm of lung
* bronchial diameter greater than adjacent segmental bronchi

Exclusion Criteria:Subject will be excluded if she or he has one of the following

* It is unable or doesn't agree to accept the follow-up process
* undergoing trial for other medications or instruments.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as bronchiectasis at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung function on the spirometry | 5 years
  forced expiratory volume at one second (FEV1) in Liter

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD,PhD, Study Director — Beijing Children's Hospital of Capital Medical University, China; Baoping Xu, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Xiaoxia Peng, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China
Locations (1):
- Beijing Children'S Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Karakoc GB, Yilmaz M, Altintas DU, Kendirli SG. Bronchiectasis: still a problem. Pediatr Pulmonol. 2001 Aug;32(2):175-8. doi: 10.1002/ppul.1104. PMID 11477735
- [Background] Munro KA, Reed PW, Joyce H, Perry D, Twiss J, Byrnes CA, Edwards EA. Do New Zealand children with non-cystic fibrosis bronchiectasis show disease progression? Pediatr Pulmonol. 2011 Feb;46(2):131-8. doi: 10.1002/ppul.21331. Epub 2010 Aug 17. PMID 20717910
- [Background] Twiss J, Stewart AW, Byrnes CA. Longitudinal pulmonary function of childhood bronchiectasis and comparison with cystic fibrosis. Thorax. 2006 May;61(5):414-8. doi: 10.1136/thx.2005.047332. Epub 2006 Feb 7. PMID 16467074
- [Background] Murray MP, Pentland JL, Hill AT. A randomised crossover trial of chest physiotherapy in non-cystic fibrosis bronchiectasis. Eur Respir J. 2009 Nov;34(5):1086-92. doi: 10.1183/09031936.00055509. Epub 2009 Jun 18. PMID 19541717
- [Background] Davies G, Wilson R. Prophylactic antibiotic treatment of bronchiectasis with azithromycin. Thorax. 2004 Jun;59(6):540-1. No abstract available. PMID 15170047
- [Background] Valery PC, Morris PS, Byrnes CA, Grimwood K, Torzillo PJ, Bauert PA, Masters IB, Diaz A, McCallum GB, Mobberley C, Tjhung I, Hare KM, Ware RS, Chang AB. Long-term azithromycin for Indigenous children with non-cystic-fibrosis bronchiectasis or chronic suppurative lung disease (Bronchiectasis Intervention Study): a multicentre, double-blind, randomised controlled trial. Lancet Respir Med. 2013 Oct;1(8):610-620. doi: 10.1016/S2213-2600(13)70185-1. Epub 2013 Sep 17. PMID 24461664
- [Background] Gaylor AS, Reilly JC. Therapy with macrolides in patients with cystic fibrosis. Pharmacotherapy. 2002 Feb;22(2):227-39. doi: 10.1592/phco.22.3.227.33544. PMID 11837560
- [Background] WANG Hao，XU Bao-ping，LIU Xiu-yun，HU Ying-hui，REN Yi-xin，SHEN Kun-ling. Clinical characteristics and follow-up of bronchiectasis in children. Chinese Journal of Practical Pediatrics, 2014;29 (12):936-939
- [Background] CHEN Jun, DUO Li-kun, WANG Xiao-feng. Clinical analysis of 22 children with bronchiectasis. J Clin Pediatr, 2012, 30(1):51-54.